CLINICAL TRIAL: NCT02810990
Title: Bosutinib Efficacy, Safety, Tolerability (BEST) Study in Elderly Chronic Myeloid Leukemia Patients Failing Front-line Treatment With Other Tyrosine Kinase Inhibitors
Brief Title: Bosutinib in Elderly Chronic Myeloid Leukemia
Acronym: BEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML1516; 2016-002216-40 (EudraCT Number)
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Chronic Myeloid Leukemia
Keywords: bosutinib; chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bosutinib treatment (Experimental)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — Bosutinib is given orally accordingly with this scheme:
  A. 200 mg OD: starting dose ("wash-in" period) at week 1 and week 2 B. 300 mg OD: from week 3 to the end of week 16
  At the end of week 12 evaluation of molecular response (BCR-ABL1 level by RT-Q-PCR).
  Bosutinib dose is then managed as follows :
  C1. if BCR-ABL1 ≤1% at week 12: 300 mg OD from week 17 to week 52 C2. if BCR-ABL1 > 1% at week 12: 400 mg OD from week 17 to week 52
  All the responsive patients who are still on Bosutinib at the end of week 52, will continue Bosutinib at the same dose (300 mg OD or 400 mg OD) for the next two years ( if tolerated and in absence of safety concerns).

SUMMARY:
The objective of the present study is to evaluate a new drug called bosutinib as it is believed that this agent may be able to predict an excellent prognosis in patients that did not obtain any benefit with other drugs before. Still, this needs to be proved and we hope this study is able to do so.

DETAILED DESCRIPTION:
Bosutinib is a potent tyrosine kinase inhibitor (TKI) active at nM concentration on BCR-ABL1 and most BCR-ABL1 mutations. Bosutinib has been approved by the FDA and the EMA for the treatment of patients with Ph+/BCR-ABL1+ chronic myeloid leukemia who fail treatment with other TKIs, first or second line. The goal of second-line treatment of CML is to achieve a response that would predict for a survival equal to, or very close to, the survival of non leukemic people, that is to say to achieve a complete cytogenetic response (CCyR) or a major molecular response (MMR). To achieve that goal, it is necessary to find and keep the right balance between activity, safety, and tolerability. There are no studies comparing TKIs in second-line. From phase 2, single-arm, studies, the reported efficacy of Bosutinib is similar to the reported efficacy of dasatinib and nilotinib. The median age of newly diagnosed CML patients is about 56 years, and at least 40% of all newly diagnosed patients are more than 60 years old. Particularly for these patients, the choice of the TKI must take into account the safety and the tolerability profile of the TKIs. The use of dasatinib and nilotinib is burdened by pleural and pulmonary complications, by infections, and by cardiovascular, thrombotic and metabolic (diabetes mellitus, dyslipidemia) complications. These complications are more frequent and more clinically relevant in the elderly. The safety and tolerability of Bosutinib has been reported in first- as well as in second- and third-line. The standard dose (500 mg once daily) is tolerated and safe, but at that dose several adverse events (AEs) limit the tolerability, require dose reduction or interruption, and affect patient quality of life, including diarrhea, nausea, vomiting, skin rash. Also an increase of AST, ALT and lipase are of concern and a cause of treatment discontinuation. On the contrary, an increased frequency of infections and of pleuro-pulmonary, cardiovascular, thrombotic, and metabolic AEs has not been reported. The reported hematologic toxicity of Bosutinib is at least as low as, or even lower than, that reported for the other TKIs, in spite of the fact that Bosutinib is a dual, BCR-ABL1 and src inhibitor. Until today, all studies of TKIs in CML have tested a fixed initial dose, providing for dose adjustment in case of toxicity (dose decrease) or in case of unsatisfactory response (dose increase). No study so far was designed to test the adaptation of the dose to the response, taking advantage of the fact that the efficacy of TKI treatment can be assessed rapidly and precisely by measuring the BCR-ABL1 transcripts level with real-time PCR (RT-PCR) in peripheral blood cells. An RT-PCR monthly for the first few months provides the best assessment of the response to treatment. We predict that a more flexible strategy of treatment (adapting the dose to the response) will result into a more convenient balance between activity and toxicity, hence into a better outcome. Based on these premises, it is proposed to test the activity, the safety, and the tolerability of Bosutinib, second-line, beginning with a low dose and adjusting subsequent doses based on molecular response, and on AEs, in a population of elderly patients. In almost all prior studies of TKIs in second- or third-line, the primary efficacy was assessed using cytogenetic response, both major and complete, at different time points. To make the results of this study comparable to the results of prior studies, the cytogenetic response will be evaluated as specified in section 5, but since the response to therapy and the evaluation of the efficacy of therapy are more and more based on molecular response, dose adaptation and efficacy evaluation will be based primarily on molecular response.

ELIGIBILITY:
Inclusion Criteria:

1. Molecular confirmed diagnosis of BCR-ABL1+ CML
2. Chronic phase CML (ELN 2013 criteria)
3. 60 years of age or older
4. Prior first-line treatment with any other TKIs
5. Intolerance to prior treatment, based on investigator and patient assessment or failure of prior treatment according to any one of the ELN 2013 criteria, as listed below

   * Non complete hematologic response (CHR) at 3 months
   * No cytogenetic response (Ph+ > 95%) at 6 months
   * Less than Partial Cytogenetic Response (PCyR) (Ph+ >35%) at 6 months
   * BCR-ABL1 > 10% at 6 months
   * Non complete CyR (CCyR) (Ph+ > 0) at 12 months
   * BCR-ABL1 > 1% at 12 months
   * Loss of CHR at any time
   * Loss of CCyR at any time
   * Confirmed loss of major molecular response (MMR) (BCR-ABL1 > 0.1%) in two consecutive tests, of which one > 1%, at any time
6. An effective form of contraception from enrolment through 30 days after the end of treatment
7. Signed written informed consent according to ICH/EU/GCP and national and local laws prior to any study procedures
8. Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Accelerated or blastic phase CML (according to ELN 2013 criteria)
2. Patients with the T315I or the V299L mutation
3. Patients previously treated with 2 TKIs or more
4. Compelled to take medications that are known to be associated with Torsades de Pointes and/or with significant QTc prolongation
5. Any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the drug
6. HBV markers positivity
7. Lack of informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-11-17 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Number of patients who are in major molecular response (MMR) | One year treatment

SECONDARY OUTCOMES:
Number of patients who obtain molecular response | At 6 and 12 months from treatment start
Number of patients discontinuing treatment for failure, adverse events or other reasons | At 12 and 36 months
Number of Adverse Events (AEs) | At 36 months
Number of patients alive | At 36 months
Number of patients on treatment at 200, 300 and 400 mg or more daily | At 6, 12 and 36 months
Number and type of BCR-ABL1 mutations | At 36 months
Patient reported quality of life | At 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Castagnetti, Study Chair — Department of Hematology, S. Orsola-Malpighi University of Bologna
Locations (45):
- Italy (45):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Fausto Castagnetti, Bologna
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Policlinico S. Orsola - Malpighi, Bologna
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - S.C. Ematologia ASO S. Croce e Carle, Cuneo
  - Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia, Ferrara
  - Policlinico di Careggi, Florence
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia, Foggia
  - IRCCS_AOU San Martino-IST-Ematologia 1-Monoblocco 11°piano- lato ponente, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia, Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - Azienda Ospedaliera "S.Gerardo", Monza
  - Azienda Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - S.C.D.U. Ematologia - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. di Ematologia con trapianto - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Ematologia - Ospedale San Carlo, Potenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Padiglione Cesalpino - I piano - Divisione di Ematologia - Ospedale S. Camillo, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - UOC Pronto Soccorso - Dipartimento Biotecnologie Cellulari Università di Roma "Sapienza", Roma
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Divisione di Ematologia - "Città della Salute e della Scienza di Torino", Torino
  - S.C. Ematologia 2 A.O. Città della Salute e della Scienza di Torino San Giovanni Battista, Torino
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari, Udine
  - Medicina Interna I - Ospedale di Circolo, Varese
  - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it